CLINICAL TRIAL: NCT06298162
Title: Assessment of Pouch Emptying With MRI After Roux-en-Y Gastric Bypass
Acronym: MRI pouch
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-1279
Record Dates: First submitted 2021-07-23; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Bariatric Surgery Candidate; Gastric Bypass; Obesity, Morbid; Pouch Emptying
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RYGB, successful weight loss (TWL >35%): TWL = total weight loss
  Interventions: Other: 2 years after RYGB, no intervention. MRI measurement. Observational.
- RYGB, unsuccessful weight loss (TWL <25%)
  Interventions: Other: 2 years after RYGB, no intervention. MRI measurement. Observational.

INTERVENTIONS:
Other: 2 years after RYGB, no intervention. MRI measurement. Observational. — no intervention. MRI measurement. Observation.

SUMMARY:
A cross-sectional observational study in which pouch emptying rate is measured with MRI in good (TWL>35%) and bad responders (TWL<25%) two years after Laparoscopic Roux-en-Y Gastric Bypass (LRYGB).

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 20 and 55 years
* Patients must be able to adhere to the study visit schedule and protocol requirements
* Patients must be able to give informed consent (IC) prior to any study procedures
* Patients who had a follow-up period up until two years after LRYGB and have successful or unsuccessful weight loss.
* Willing to be informed about incidental findings of pathology and approving of reporting this to their general physician

Exclusion Criteria:

* Diabetes Mellitus
* Menopausal
* Gastrointestinal problems, gastric or intestinal diseases
* Drug or alcohol addiction
* Inability to stop smoking during the overnight fasting period
* Pregnant or lactating
* Having an intolerance or allergy for one of the components of the test product
* Inability to stop medications that affect gastrointestinal emptying like antisecretory drugs, narcotics and prokinetic agents
* Inability to stop medication that affects the motility of the upper gastrointestinal tract (anti-cholinergic drugs, prokinetics, theophylline, calcium blocking agents, opioids)
* Having a contra-indication to MRI scanning (including, but not limited to):

  * Pacemakers and defibrillators
  * Intraorbital or intraocular metallic fragments
  * Ferromagnetic implants

Ages: 20 Years to 55 Years | Sex: Female
Age Groups: Adult
Study Population: RYGB, with succesful (>35%) or unsuccesful (<25%) weight loss
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Pouch emptying rate measured with MRI | Two years after LRYGB

SECONDARY OUTCOMES:
subjective ratings of fullness | Two years after LRYGB
  subjective ratings of fullness will be measured an a 100-unit Visual Analogue Scale
subjective ratings of wellbeing | Two years after LRYGB
  subjective ratings of wellbeing will be measured an a 100-unit Visual Analogue Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Yonta Burgh, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided